CLINICAL TRIAL: NCT03596801
Title: Phase I Placebo-Controlled Study of the Infectivity, Safety and Immunogenicity of a Single Dose of a Recombinant Live-attenuated Respiratory Syncytial Virus Vaccine, RSV 6120/∆NS1, Lot RSV#018A, or RSV 6120/F1/G2/∆NS1, Lot RSV#016A, Delivered as Nose Drops to RSV-seropositive Children 12 to 59 Months of Age and RSV-seronegative Infants and Children 6 to 24 Months of Age
Brief Title: Evaluating the Infectivity, Safety and Immunogenicity of Respiratory Syncytial Virus Vaccines, RSV 6120/∆NS1 and RSV 6120/F1/G2/∆NS1, in RSV-Seropositive Children and RSV-Seronegative Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 330
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: RSV 6120/∆NS1 Vaccine (Experimental): Healthy RSV-seropositive children greater than or equal to 12 months to less than 60 months will receive a single dose of 10^6.0 plaque-forming units (PFUs) of RSV 6120/∆NS1 vaccine at Day 0.
  Interventions: Biological: RSV 6120/∆NS1
- Group 1: RSV 6120/F1/G2/∆NS1 Vaccine (Experimental): Healthy RSV-seropositive children greater than or equal to 12 months to less than 60 months will receive a single dose of 10^5.8 PFUs of RSV 6120/F1/G2/∆NS1 vaccine at Day 0.
  Interventions: Biological: RSV 6120/F1/G2/∆NS1
- Group 1: Placebo (Placebo Comparator): Healthy RSV-seropositive children greater than or equal to 12 months to less than 60 months will receive a single dose of placebo at Day 0.
  Interventions: Biological: Placebo
- Group 2: RSV 6120/∆NS1 Vaccine (Experimental): Healthy RSV-seronegative infants and children greater than or equal to 6 months to less than 25 months will receive a single dose of 10^5.0 PFUs of RSV 6120/∆NS1 vaccine at Day 0.
  Interventions: Biological: RSV 6120/∆NS1
- Group 2: RSV 6120/F1/G2/∆NS1 (Experimental): Healthy RSV-seronegative infants and children greater than or equal to 6 months to less than 25 months will receive a single dose of 10^5.0 PFUs of RSV 6120/F1/G2/∆NS1 vaccine at Day 0.
  Interventions: Biological: RSV 6120/F1/G2/∆NS1
- Group 2: Placebo (Placebo Comparator): Healthy RSV-seronegative infants and children greater than or equal to 6 months to less than 25 months will receive a single dose of placebo at Day 0.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV 6120/∆NS1 — Delivered as nose drops
  Arms: Group 1: RSV 6120/∆NS1 Vaccine; Group 2: RSV 6120/∆NS1 Vaccine
Biological: RSV 6120/F1/G2/∆NS1 — Delivered as nose drops
  Arms: Group 1: RSV 6120/F1/G2/∆NS1 Vaccine; Group 2: RSV 6120/F1/G2/∆NS1
Biological: Placebo — Delivered as nose drops
  Arms: Group 1: Placebo; Group 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the infectivity, safety, and immunogenicity of a single dose of recombinant, live-attenuated respiratory syncytial virus (RSV) vaccines (RSV 6120/∆NS1 or RSV 6120/F1/G2/∆NS1) in RSV-seropositive children 12 to 59 months of age and RSV-seronegative infants and children 6 to 24 months of age.

DETAILED DESCRIPTION:
This study will evaluate the infectivity, safety, and immunogenicity of a single dose of recombinant, live-attenuated respiratory syncytial virus (RSV) vaccines (RSV 6120/∆NS1 or RSV 6120/F1/G2/∆NS1) in RSV-seropositive children 12 to 59 months of age and RSV-seronegative infants and children 6 to 24 months of age.

The vaccines will be evaluated in a stepwise fashion beginning with RSV-seropositive children (Group 1) and proceeding sequentially in RSV-seronegative infants and children (Group 2). In each group, participants will be randomly assigned to receive a single dose of RSV 6120/∆NS1, RSV 6120/F1/G2/∆NS1, or placebo at Day 0.

Participants will be enrolled in the study between April 1 and October 31, outside of the RSV season. Group 1 participants will be followed for 28 days after inoculation, and Group 2 participants will remain on the study until they complete the post-RSV season visit between April 1 and April 30 in the calendar year following enrollment. The expected duration of the initial study is 28 days for Group 1 participants and between 6 and 13 months for Group 2 participants, depending upon time of enrollment.

Study visits for all participants may include clinical assessments, blood collection, and nasal washes. Additionally, participants' parents or guardians will be contacted by study staff at various times during the study to monitor participants' health.

ELIGIBILITY:
INCLUSION CRITERIA FOR RSV-SEROPOSITIVE CHILDREN

* Greater than or equal to 12 months of age and less than 60 months of age at the time of inoculation
* Screening serum specimen for RSV-neutralizing antibody is obtained within the calendar year of inoculation
* Seropositive for RSV antibody, defined as serum RSV-neutralizing antibody titer greater than or equal to 1:40
* Pre-inoculation serum sample for RSV-neutralizing antibody specimen is obtained no more than 56 days prior to inoculation
* In good health based on review of the medical record, history, and physical examination (PE) at the time of inoculation
* Received routine immunizations appropriate for age based on the Advisory Committee on Immunization Practices (ACIP) Recommended Immunization Schedule for Children and Adolescents Aged 18 Years or Younger
* Growing normally for age as demonstrated on a standard growth chart and has a current height and weight above the 3rd percentile for age
* Expected to be available for the duration of the study
* Parent/guardian is willing and able to provide written informed consent

EXCLUSION CRITERIA FOR RSV-SEROPOSITIVE CHILDREN

* Born at less than 34 weeks gestation
* Maternal history of positive human immunodeficiency virus (HIV) test
* Evidence of chronic disease
* Known or suspected impairment of immune function
* Bone marrow/solid organ transplant recipient
* Major congenital malformations, including congenital cleft palate or cytogenetic abnormalities
* Suspected or documented developmental disorder, delay, or other developmental problem
* Cardiac abnormality requiring treatment
* Lung disease or reactive airway disease
* More than one episode of wheezing in the first year of life
* Wheezing episode or received bronchodilator therapy within the past 12 months
* Wheezing episode or received bronchodilator therapy after the age of 12 months
* Previous receipt of supplemental oxygen therapy in a home setting
* Previous receipt of an investigational RSV vaccine
* Previous receipt or planned administration of anti-RSV antibody product including ribavirin, RSV Ig or RSV mAb
* Previous receipt of immunoglobulin or any antibody products within the past 6 months
* Previous receipt of any other blood products within the past 6 months
* Previous anaphylactic reaction
* Previous vaccine-associated adverse reaction that was Grade 3 or above
* Known hypersensitivity to any vaccine component
* Member of a household that contains an infant who is less than 12 months of age at the date of inoculation through the 10th day after inoculation
* Member of a household that, at the date of inoculation through the 10th day after inoculation, contains an immunocompromised individual including but not limited to:

  * a person who is HIV-infected
  * a person who has received chemotherapy within the 12 months prior to enrollment
  * a person receiving immunosuppressant agents
  * a person living with a solid organ or bone marrow transplant
* Will attend a daycare facility that does not separate children by age and contains an infant who is less than 12 months of age at the date of inoculation through the 10th day after inoculation
* Receipt of any of the following prior to enrollment:

  * any inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior, or
  * salicylate (aspirin) or salicylate-containing products within the past 28 days
* Scheduled administration of any of the following after planned inoculation:

  * inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus within the 28 days after, or
  * another investigational vaccine or investigational drug within the 28 days after
* Receipt of any of the following medications within 3 days of study enrollment:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medications except the permitted concomitant medications listed in the protocol
* Any of the following events at the time of enrollment:

  * fever (temporal or rectal temperature of greater than or equal to 100.4°F), or
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis) or
  * nasal congestion significant enough to interfere with successful inoculation, or
  * otitis media

INCLUSION CRITERIA FOR RSV-SERONEGATIVE INFANTS & CHILDREN

* Greater than or equal to 6 months of age and less than 25 months of age at the time of inoculation
* Screening and pre-inoculation serum specimens for RSV-neutralizing antibody are obtained no more than 42 days prior to inoculation
* Seronegative for RSV antibody, defined as serum RSV-neutralizing antibody titer less than 1:40
* In good health based on review of the medical record, history, and PE at the time of inoculation
* Received routine immunizations appropriate for age based on the ACIP Recommended Immunization Schedule for Children and Adolescents Aged 18 Years or Younger
* Growing normally for age as demonstrated on a standard growth chart, AND

  * If less than 1 year of age: has a current height and weight above the 5th percentile for age
  * If greater than or equal to 1 year of age: has a current height and weight above the 3rd percentile for age
* Expected to be available for the duration of the study
* Parent/guardian is willing and able to provide written informed consent

EXCLUSION CRITERIA FOR RSV-SERONEGATIVE INFANTS & CHILDREN

* Born at less than 34 weeks gestation
* Born at less than 37 weeks gestation, and at the date of inoculation less than 1 year of age
* Maternal history of a positive HIV test
* Evidence of chronic disease
* Known or suspected infection or impairment of immunological functions
* Bone marrow/solid organ transplant recipient
* Major congenital malformations, including congenital cleft palate or cytogenetic abnormalities
* Suspected or documented developmental disorder, delay, or other developmental problem
* Cardiac abnormality requiring treatment
* Lung disease or reactive airway disease
* More than one episode of wheezing in the first year of life
* Wheezing episode or received bronchodilator therapy within the past 12 months
* Wheezing episode or received bronchodilator therapy after the age of 12 months
* Previous receipt of supplemental oxygen therapy in a home setting
* Previous receipt of an investigational RSV vaccine
* Previous receipt or planned administration of anti-RSV antibody product including ribavirin, RSV Ig, or RSV mAb
* Previous receipt of immunoglobulin or any antibody products within the past 6 months
* Previous receipt of any blood products within the past 6 months
* Previous anaphylactic reaction
* Previous vaccine-associated adverse reaction that was Grade 3 or above
* Known hypersensitivity to any study product component
* Member of a household that contains an infant who is less than 6 months of age at the date of inoculation through the 28th day after inoculation
* Member of a household that, at the date of inoculation through the 28th day after inoculation, contains an immunocompromised individual including but not limited to:

  * a person who is HIV-infected
  * a person who has received chemotherapy within the 12 months prior to enrollment
  * a person receiving immunosuppressant agents
  * a person living with a solid organ or bone marrow transplant
* Attends a daycare facility that does not separate children by age and contains an infant less than 6 months of age at the date of inoculation through the 28th day after inoculation
* Receipt of any of the following prior to enrollment:

  * any inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior, or
  * salicylate (aspirin) or salicylate-containing products within the past 28 days
* Scheduled administration of any of the following after planned inoculation

  * inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus within the 28 days after, or
  * another investigational vaccine or investigational drug within the 56 days after
* Receipt of any of the following medications within 3 days of study enrollment:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medications except the permitted concomitant medications listed below
  * Permitted concomitant medications (prescription or non-prescription) include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) cutaneous (topical) steroids, topical antibiotics, and topical antifungal agents.
* Any of the following events at the time of enrollment:

  * fever (temporal or rectal temperature of greater than or equal to 100.4°F), or
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis) or
  * nasal congestion significant enough to interfere with successful inoculation, or
  * otitis media

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Grades of study product-related solicited adverse events (AEs) (RSV-seropositive participants) | Measured through Day 10
  Graded using the protocol-defined grading system
Grades of study product-related solicited AEs (RSV-seronegative participants) | Measured through Day 28
  Graded using the protocol-defined grading system
Grades of study product-related unsolicited AEs (RSV-seropositive participants) | Measured through Day 10
  Graded using the protocol-defined grading system
Grades of study product-related unsolicited AEs (RSV-seronegative participants) | Measured through Day 28
  Graded using the protocol-defined grading system
Grades of study product-related serious adverse events (SAEs) (RSV-seropositive participants) | Measured through Day 28
  Graded using the protocol-defined grading system
Grades of study product-related SAEs (RSV-seronegative participants) | Measured through Day 56
  Graded using the protocol-defined grading system
Frequency of infection with RSV (RSV-seropositive participants) | Measured through Day 28
  Defined as 1) vaccine virus identified in nasal wash (a binary outcome based on nasal washes done throughout the study period; Day 0 nasal wash will be counted as baseline) or 2) a greater than or equal to 4-fold rise in serum RSV neutralizing antibody titer or serum RSV F (IgG) titer
Frequency of infection with RSV (RSV-seronegative participants) | Measured through Day 56
  Defined as 1) vaccine virus identified in nasal wash (a binary outcome based on nasal washes done throughout the study period; Day 0 nasal wash will be counted as baseline) or 2) a greater than or equal to 4-fold rise in serum RSV neutralizing antibody titer or serum RSV F (IgG) titer
Peak titer of vaccine virus shed (RSV-seropositive participants) | Measured through Day 10
  Based on laboratory evaluations
Peak titer of vaccine virus shed (RSV-seronegative participants) | Measured through Day 28
  Based on laboratory evaluations
Duration of virus shedding in nasal washes (RSV-seropositive participants) | Measured through Day 10
  As determined by a) culture and b) reverse transcription polymerase chain reaction (rRT-PCR)
Duration of virus shedding in nasal washes (RSV-seronegative participants) | Measured through Day 28
  As determined by a) culture and b) rRT-PCR
Frequency of a greater than or equal to 4-fold rise in RSV-neutralizing antibody titer (RSV-seropositive participants) | Measured through Day 28
  Based on laboratory evaluations
Frequency of a greater than or equal to 4-fold rise in RSV-neutralizing antibody titer (RSV-seronegative participants) | Measured through Day 56
  Based on laboratory evaluations
Frequency of a greater than or equal to 4-fold rise in immunoglobulin G (IgG) antibody responses to RSV F glycoprotein (RSV-seropositive participants) | Measured through Day 28
  As determined by ELISA
Frequency of a greater than or equal to 4-fold rise in IgG antibody responses to RSV F glycoprotein (RSV-seronegative participants) | Measured through Day 56
  As determined by ELISA

SECONDARY OUTCOMES:
Frequency of symptomatic, medically attended respiratory and febrile illness in the RSV-seronegative (group 2) vaccine and placebo recipients who experience natural infection with wt RSV during the RSV season | Measured through participants' last study visit at 6 to 13 months, depending on when participants enroll in the study
  Based on laboratory evaluations
Severity of symptomatic, medically attended respiratory and febrile illness in the RSV-seronegative (group 2) vaccine and placebo recipients who experience natural infection with wt RSV during the RSV season | Measured through participants' last study visit at 6 to 13 months, depending on when participants enroll in the study
  Based on laboratory evaluations
Frequency of antibody responses in the RSV-seronegative vaccine and placebo recipients who experience natural infection with wt RSV during the RSV season | Measured through participants' last study visit at 6 to 13 months, depending on when participants enroll in the study
  Based on laboratory evaluations
Measurement of mucosal antibody titers to vaccine | Measured through participants' last study visit at 6 to 13 months, depending on when participants enroll in the study
  Assessed in nasal wash or nasosorption samples

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health (JHSPH)
Locations (1):
- Johns Hopkins University Center for Immunization Research, Baltimore, Maryland, United States